CLINICAL TRIAL: NCT02891421
Title: Effects of Equine Assisted Activities on PTSD Symptoms, Coping Self-efficacy, Emotion Regulation, and Social Engagement in U.S. Military Veterans
Brief Title: Therapeutic Horsemanship in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Harry S. Truman Memorial Veterans' Hospital (U.S. Federal Agency); Horses and Humans Research Foundation (Unknown)
Responsible Party: Principal Investigator, Rebecca Johnson, Prinicipal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1207664-1
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Post Traumatic Stress Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic | interventions — Standard of Care

ARMS (2):
- Therapeutic Horseback Riding (Other): Therapeutic Horseback Riding: Veterans were matched to a horse by the instructor and occupational therapist for best fit and the same horse was ridden each week
  Interventions: Behavioral: Therapeutic Horseback Riding
- Standard Care (Other): Participants received standard care.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Therapeutic Horseback Riding — Veterans were matched to a horse for best fit and the same horse was ridden each week. The warm-up exercises involved various repeated physical movements while the horse was walking or standing steady, such as head rotations, lifting arms, rotating ankles, flexing toes. The exercises began with riding at a walk during the early weeks, learning reining skills and riding positions, and progressed to light trotting. Veteran participants were able to build on skill sets related to grooming, tacking, mounting, and riding that were introduced in prior weeks. Skill progression was based on individual abilities and safety as determined by certified riding instructor and occupational therapist.
  Arms: Therapeutic Horseback Riding
Other: Standard Care — Standard Care: Participants received standard care
  Arms: Standard Care

SUMMARY:
The project partnered with U.S. military veterans with a premier accredited therapeutic riding center for six weeks. The veterans interacted with horses by grooming and learning about them, as well as riding them for one hour per week during which they gained a variety of skills. We hoped the veterans would experience a reduction in Post Traumatic Stress Disorder (PTSD) symptoms, depression, and loneliness, while improving their social and emotional health and self-efficacy.

DETAILED DESCRIPTION:
Large numbers of post-deployed U.S. veterans diagnosed with Post Traumatic Stress Disorder (PTSD) and/or Traumatic Brain Injury make effective interventions urgent, to reduce symptoms and increase veterans' coping. PTSD includes anxiety, flashbacks, and emotional numbing. Symptoms expand health care costs for stress-related illnesses making veterans' civilian life difficult.

The proposed study used a randomized experimental design with repeated measures and waitlist control group testing the efficacy of a 6-week human-horse interaction and systematic therapeutic horseback riding program in: decreasing PTSD symptoms, increasing coping self efficacy, emotion regulation, and social engagement. The Riding Group spent one hour weekly interacting with and riding the same horse at one of two PATH-accredited riding centers in Mid-Missouri supervised by an Occupational Therapist, Profession Association of Therapeutic Horsemanship (PATH) International-certified instructor, leader and side walkers as needed. Riding was directed by a systematic lesson plan. Data collection occured at baseline, 3 weeks, and 6 weeks. The Control Group was assessed at the same intervals and again 3 weeks and 6 weeks after joining the Riding Group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Veterans, left active military service (not serving in reserve units.)
* Diagnosed with Post Traumatic Stress Disorder/Traumatic Brain Injury or both according to ICD-9 diagnostic codes.
* Weight less than 220 pounds.
* Able to walk at least 25 feet without the assistance of a person (but potentially with assistive devices).
* Willing to interact with and ride a horse.
* Have not ridden a horse in the past year.
* Care Provider assent

Exclusion Criteria:

* Age less than 18 years
* Veterans in active military service (including reserve units).
* No diagnosis of PTSD/TBI or both according to ICD-9 diagnostic codes.
* Weight greater than 221 pounds.
* Unable to walk at least 25 feet without the assistance of a person (but potentially with assistive devices.)
* Unwilling to interact with and ride a horse.
* Have been riding a horse in the past year.
* Care Provider unwilling to provide assent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Coping Self-Efficacy Scale (CSES) | Day 1, 3 weeks and 6 weeks
  26 item, 11 point analog scale
Change in Post-Traumatic Stress Disorder Checklist-Military Version (PCL-M) | Day 1, 3 weeks and 6 weeks
  17 item, 5 point scale

SECONDARY OUTCOMES:
Change in Social and Emotional Loneliness Scale for Adults (SELSA) scale | Day 1, 3 weeks and 6 weeks
  15 item, 7 point Likert-type scale.
Change in Difficulties in Emotion Regulation Scale (DERS) | Day 1, 3 weeks and 6 weeks
  36 item, 5 point Likert-type scale

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Johnson, PhD, Principal Investigator — University of Missouri-Columbia

REFERENCES:
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720
- [Background] Brewin CR, Andrews B, Valentine JD. Meta-analysis of risk factors for posttraumatic stress disorder in trauma-exposed adults. J Consult Clin Psychol. 2000 Oct;68(5):748-66. doi: 10.1037//0022-006x.68.5.748. PMID 11068961
- [Background] Hakanson M, Moller M, Lindstrom I, Mattsson B. The horse as the healer-a study of riding in patients with back pain. J Bodyw Mov Ther. 2009 Jan;13(1):43-52. doi: 10.1016/j.jbmt.2007.06.002. Epub 2007 Aug 24. PMID 19118792
- [Background] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750